CLINICAL TRIAL: NCT00587691
Title: An Open-Label, Dose-Escalation Study of T Cell Vaccine in Multiple Sclerosis
Brief Title: Dose-Escalation Study of T Cell Vaccine in Multiple Sclerosis
Acronym: DES
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Opexa Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000-03
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Secondary Progressive
Keywords: Tovaxin; TCV; Autologous
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dose Level 1 (Experimental): 6-9 million MRTC
  Interventions: Biological: Tovaxin Autologous T Cell Vaccine
- Dose Level 2 (Experimental): 30-45 million MRTC
  Interventions: Biological: Tovaxin Autologous T Cell Vaccine
- Dose Level 3 (Experimental): 60-90 million MRTC
  Interventions: Biological: Tovaxin Autologous T Cell Vaccine

INTERVENTIONS:
Biological: Tovaxin Autologous T Cell Vaccine — Primary Series (x1): 4 subcutaneous injections (wks 0, 4, 12 and 20 with 52 week evaluable period.
  Retreatment Series (x3): 3 subcutaneous injections (wks 0, 4, and 8) with 26-week evaluable periods.
  Retreatment Series (x3): 5 subcutaneous injections (wks 0, 8, 26, 24 and 32) with 52-week evaluable periods.

SUMMARY:
The purpose of the study is 1) to study the safety and tolerability of escalating doses of myelin peptide reactive T cells in MS patients and 2) to study the clinical effectiveness of T Cell Vaccine ion the clinical course of MS.

DETAILED DESCRIPTION:
The principle of TCV is similar to that of traditional microbial vaccination where attenuated infectious agents are used to stimulate protective immune responses. Because pathogentic autoreactive T cells are viewed as pathogens in T cell-mediated autoimmune diseases, they can be used, as a vaccine to prevent and treat the diseases in which they are able to induce.

ELIGIBILITY:
Inclusion Criteria:

* Stable MS disease within 30 days prior to enrollment
* EDSS Score between 2 and 8 inclusively
* Failed to respond to or cannot tolerate at least 1 or more of the currently approved drugs for MS.

Exclusion Criteria:

* Women who are pregnant or breast-feeding or who plan to become pregnant during the study
* Has taken immunomodulating drugs within 60 days prior to screening
* HIV positive

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2002-07; Primary Completion 2007-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety and tolerability | Yearly Intervals

SECONDARY OUTCOMES:
To assess changes in EDSS Scores | Yearly Intervals
To assess changes in the myelin-reactive profile in the blood | Yearly Intervals
To assess changes in the frequency of MS relapses | Yearly Intervals

CONTACTS AND LOCATIONS:
Overall Officials: Jaye Thompson, PhD, Study Director — Opexa Therapeutics
Locations (2):
- United States (2):
  - Bellaire Neurology, Bellaire, Texas
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang J. T-cell vaccination in multiple sclerosis: immunoregulatory mechanism and prospects for therapy. Crit Rev Immunol. 2001;21(1-3):41-55. PMID 11642613
- [Background] Zhang J. T-cell vaccination for autoimmune diseases: immunologic lessons and clinical experience in multiple sclerosis. Expert Rev Vaccines. 2002 Oct;1(3):285-92. doi: 10.1586/14760584.1.3.285. PMID 12901569
- [Background] Zhang JZ, Rivera VM, Tejada-Simon MV, Yang D, Hong J, Li S, Haykal H, Killian J, Zang YC. T cell vaccination in multiple sclerosis: results of a preliminary study. J Neurol. 2002 Feb;249(2):212-8. doi: 10.1007/pl00007867. PMID 11985389